CLINICAL TRIAL: NCT05939440
Title: Proactive Costs of Care Interventions to Decrease Financial Toxicity in Cancer Patients.
Brief Title: Interventions to Decrease Financial Toxicity
Acronym: P-COC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: O'Neal Comprehensive Cancer Center at UAB (Unknown)
Responsible Party: Principal Investigator, Maria Pisu, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UAB2198
Record Dates: First submitted 2023-06-09; First posted 2023-07-11 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cancer, Breast; Cancer Colorectal; Cancer, Ovarian; Cervical Cancer; Uterine Cancer; Vulvar Cancer
Keywords: financial toxicity; financial distress; costs of care
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms; Vulvar Neoplasms; Financial Stress | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective trial
Who Masked: Outcomes Assessor
Masking Description: Assessors who conduct surveys are blind to study assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proactive Cost of Care (P-COC) intervention (Experimental): One time session with trained educator to review:
  1. Cost Information Flyer: Anticipated out of pocket costs flyer by cancer type and stage
  2. Cost Tracking workbook: Out-of-pocket cost tracker Participants also review a "Insurance, Employment, and Financial Assistance flyer" Participants will be reminded to track their costs once a month through an automated text message or e-mail based on patient preference.
  Participants also receive an existing patient pamphlet "Patient and Family Guide"
  Interventions: Other: Proactive Cost of Care (P-COC) intervention
- Usual Care (Active Comparator): Participants receive an existing patient pamphlet "Patient and Family Guide"
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Proactive Cost of Care (P-COC) intervention — As in Arm description
  Arms: Proactive Cost of Care (P-COC) intervention
Other: Usual Care — As in Arm description
  Arms: Usual Care

SUMMARY:
Financial distress affects 30-70% of cancer patients and describes the burden that patients experience due to the costs of care (CoC). One reason may be because patients lack the appropriate information on CoC that would help them better plan for and manage their CoC. Therefore, the investigators plan to test a Proactive CoC intervention which includes a discussion with a trained educator on CoC information and a Cost Tracking tool to help patients deal with their CoC.

DETAILED DESCRIPTION:
The investigators will recruit 60 patients diagnosed with gynecologic (ovarian, uterine, cervical, or vulvar cancer), breast or colorectal cancer who are starting a new line of treatment at the O'Neal Comprehensive Cancer Center. Participants will be randomized to Proactive CoC intervention versus Usual Care. Usual Care consists of the current care processes at the cancer center where information on CoC and financial assistance are only provided once a financial need is identified. The main goal is to compare the change in financial distress from baseline to 6 months to see if patients who received any of the Proactive CoC intervention have improved financial distress compared to those in Usual Care.

All participants will complete two main surveys at 0 and 6 months that will ask questions to measure the study outcomes, self-efficacy (patient reported confidence managing certain situations, such as dealing with CoC), depression, anxiety, and insurance knowledge. Participants randomized to any of the Proactive CoC intervention groups will complete three additional phone interviews at 2, 4, and 6 months to check how participants utilized the materials, reasons why they have or have not, and what sections were helpful or not. This study is important to determine whether the Proactive CoC intervention can be successfully delivered, whether the intervention is useful to help patients decrease financial distress, and to inform the design of a future larger study that will include different cancer types and health systems.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ovarian cancer (i.e., stage II-IV epithelial histology receiving surgery and chemotherapy), or newly diagnosed cervical cancer (i.e., locally advanced stage IB3-IVA receiving chemoradiation), or newly diagnosed uterine cancer (i.e., high-risk histology likely to receive chemotherapy; serous/clear cell), or newly diagnosed stage I-III breast cancer (i.e., high-risk histology), or newly diagnosed stage III-IV Colorectal Cancer
* Receiving systemic therapy or radiation at University of Alabama at Birmingham O'Neal Comprehensive Cancer Center
* With health insurance coverage
* With reliable access to a phone, mobile device, or Internet

Exclusion Criteria:

* Unable to read English
* Does not agree to complete surveys

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Financial Distress | Baseline
  FD measured using the Comprehensive Score for Financial Toxicity (COST) (12 items) The score ranges from 0 to 44 with lower scores indicating worse financial distress. A Score <26 indicates financial distress is present.
Financial Distress | 6 months
  FD measured using the Comprehensive Score for Financial Toxicity (COST) (12 items). The score ranges from 0 to 44 with lower scores indicating worse financial distress. A Score <26 indicates financial distress is present.

SECONDARY OUTCOMES:
Self Efficacy | Baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy Scale (10 items). Questions ask patients to rate their level of confidence managing situations, problems, and events related to dealing with costs of care. Responses are on a scale of 1 "I am not at all confident" to 5 "I am very confident." Self-efficacy is scored by converting raw scores into a T-score resulting in a standardized score with a mean of 50 and a standard deviation of 10.A higher score indicates more self-efficacy.
Self Efficacy | 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy Scale (10 items). Questions ask patients to rate their level of confidence managing situations, problems, and events related to dealing with costs of care. Responses are on a scale of 1 "I am not at all confident" to 5 "I am very confident." Self-efficacy is scored by converting raw scores into a T-score resulting in a standardized score with a mean of 50 and a standard deviation of 10. A higher score indicates more self-efficacy.
Depression | Baseline
  Patient Health Questionnaire (PHQ-9). Responses range from 0 "Not at all" to 3 "Nearly every day". Cut points of 5, 10, 15, and 20 are used for mild, moderate, moderately severe, and severe depression. Investigators will dichotomize into mild vs. at least moderate depression.
Depression | 6 months
  Patient Health Questionnaire (PHQ-9). Responses range from 0 "Not at all" to 3 "Nearly every day". Cut points of 5, 10, 15, and 20 are used for mild, moderate, moderately severe, and severe depression. Investigators will dichotomize into mild vs. at least moderate depression.
Anxiety | Baseline
  General Anxiety Disorder (GAD-7). Responses range from 0 "Not at all" to 3 "Nearly every day". Cut points of 5, 10, and 15 are used for mild, moderate, and severe anxiety. Responses will be dichotomized into mild vs. at least moderate anxiety.
Anxiety | 6 months
  General Anxiety Disorder (GAD-7). Responses range from 0 "Not at all" to 3 "Nearly every day". Cut points of 5, 10, and 15 are used for mild, moderate, and severe anxiety. Responses will be dichotomized into mild vs. at least moderate anxiety.
Stress | Baseline
  Weekly Stress Inventory - Short Form (WSI-SF). 25-item self-report scale that measures the number of minor stressors that occur in one week. Individual items are scored on an 8-point Likert scale. Two scores are obtained, the event score (WSI-SFE), which ranges from 0-25, and the impact score (WSI-SFI), which ranges from 0-175. A higher event score indicates more stressors and a higher impact score indicates a higher impact from these stressors.
Stress | 6 months
  Weekly Stress Inventory - Short Form (WSI-SF). 25-item self-report scale that measures the number of minor stressors that occur in one week. Individual items are scored on an 8-point Likert scale. Two scores are obtained, the event score (WSI-SFE), which ranges from 0-25, and the impact score (WSI-SFI), which ranges from 0-175. A higher event score indicates more stressors and a higher impact score indicates a higher impact from these stressors.

OTHER OUTCOMES:
Health Insurance Literacy | Baseline
  Health insurance literacy measure (HILM) measures the ability for individuals to choose and use private health insurance. Given the goals of our intervention to help patients use rather than choose health insurance, questions included those assessing confidence using insurance (5 questions) and being proactive when using health insurance (4 questions). Each question is assessed on a scale from 1 (not at all confident) to 4 (very confident). Within each domain (confidence using insurance, being proactive when using health insurance), a higher score indicates more confidence or being more proactive, respectively.
Health Insurance Literacy | 6 months
  Health insurance literacy measure (HILM) measures the ability for individuals to choose and use private health insurance. Given the goals of our intervention to help patients use rather than choose health insurance, questions included those assessing confidence using insurance (5 questions) and being proactive when using health insurance (4 questions). Each question is assessed on a scale from 1 (not at all confident) to 4 (very confident). Within each domain (confidence using insurance, being proactive when using health insurance), a higher score indicates more confidence or being more proactive, respectively.
Health Insurance Knowledge | Baseline
  Kaiser Health Insurance Knowledge Survey - 10 items - Scores range from 0-10 based on number of correct responses.
Health Insurance Knowledge | 6 months
  Kaiser Health Insurance Knowledge Survey - 10 items - Scores range from 0-10 based on number of correct responses.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pisu, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- O'Neal Comprehensive Cancer Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No